CLINICAL TRIAL: NCT02670395
Title: A Double Blind, Placebo-Controlled, Randomized, Single Ascending Dose Study to Investigate the Safety, Tolerability, Food Effect, and Pharmacokinetics of JNJ-54416076 in Healthy Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Food Effect, and Pharmacokinetics of JNJ-54416076 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108105; 54416076EDI1001 (Other: Janssen Research & Development, LLC); 2015-004162-29 (EudraCT Number)
Record Dates: First submitted 2016-01-29; First posted 2016-02-01 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54416076; Ascending Dose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- JNJ-54416076 (Experimental): Participants will receive single dose of JNJ-54416076 (in ascending dose) in Part 1 and 2 doses of JNJ-54416076 (one dose in the fasted state and an identical dose in the fed state) in Part 2. The dose selected for Part 2 will be selected based on the preliminary safety and PK data in Part 1.
  Interventions: Drug: JNJ-54416076
- Placebo (Experimental): Participants will receive single dose of placebo in Part 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-54416076 — JNJ-54416076 suspension will be administered orally.
  Arms: JNJ-54416076
Drug: Placebo — Placebo solution will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of JNJ-54416076 and any associated metabolite(s) (in Part 1) and safety, tolerability and PK of JNJ-54416076 when co administered with food compared to administration in fasting condition (in Part 2).

DETAILED DESCRIPTION:
This is a Phase 1, single-center, first-in-human study consists of 2 parts : a) Single Ascending Dose part and b) PK-Food Effect part. Part 1 is a randomized (the study medication is assigned by chance), double-blind (neither the Investigator nor the participant know the treatment), sequential cohort, single ascending oral dose study. Part 1 will assess the safety, tolerability, and PK of single ascending doses of JNJ-54416076 in healthy male participants. It will consist of 8 cohorts of 8 healthy participants. Within each cohort, 6 participants will be randomly assigned to JNJ-54416076 treatment, and 2 participants will be randomly assigned to placebo treatment. The total study duration for each participant in Part 1 will be up to approximately 5 weeks. Part 2 is a randomized, open-label (all people know the identity of the intervention), 2-period crossover study. Part 2 will assess the effect of food on the pharmacokinetics of JNJ-54416076. Each participant in Part 2 will receive 2 doses of JNJ-54416076 (one dose in the fasted state and an identical dose in the fed state). The dose selected for Part 2 will be selected based on the preliminary safety and PK data in Part 1. The total study duration for each participant in Part 2 will be up to approximately 7 weeks. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 29.9 kilogram per square meter (kg/m^2) (inclusive) and body weight greater than or equal to (>=) 50 kg
* Healthy on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and 12-lead electrocardiogram (ECG) performed at Screening. If any of the results (except for liver function and hematology tests results as defined in the protocol) are abnormal, the participant may be included only if the investigator judges that the abnormalities or deviations from normal are not clinically significant. This determination must be recorded in the participants source documents and initialed by the investigator
* Blood pressure (after the participant is sitting for 5 minutes) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and between 50 and 90 mmHg diastolic, inclusive
* Men must agree to use condoms (including men who have had vasectomies) even if their partner is pregnant (this is to ensure that the fetus is not exposed to the study drug through vaginal absorption) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug. Male participants should encourage their female partner to use an effective method (example, prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, and contraceptive patch) of contraception in addition to the condom used by the male study participant
* 18 and 45 years of age, inclusive

Exclusion Criteria:

* History of, or currently active, significant illness or medical disorders, including (but not limited to) cardiovascular disease (including cardiac arrhythmias, myocardial infarction, stroke, peripheral vascular disease), endocrine or metabolic disease (example, hyper/hypo-thyroidism), hematological disease (example, von Willebrand's disease or other bleeding disorders), respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmologic disorders (including retinal disorders or cataracts), neoplastic disease, skin disorder, renal disorder, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History of Gilbert's disease, Dubin-Johnson or Rotor syndrome, or any family history of liver or gallbladder disease that may suggest an underlying genetic disorder
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT), bilirubin levels (indirect, or direct), or alkaline phosphtase above the upper limit of normal of the clinical laboratory's reference range at Screening or at Day -1
* Hemoglobin, hematocrit, or red blood cell count below the lower limit of normal of the clinical laboratory's reference range at Screening. On Day -1, if participants have hemoglobin, hematocrit, or red blood cell count below the lower limit of normal of the clinical laboratory's reference range, the participants may be included if the investigator judges that the abnormalities or deviations from the reference range are not clinically significant
* History of cholecystectomy or gallbladder disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up visit (7 to 10 days after last study procedure)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time To Reach The Maximum Observed Concentration (Tmax) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post-dose on Day 1
  Tmax is the actual sampling time to reach the maximum observed concentration.
Area Under the Concentration Versus Time Curve (AUC) From Time of Administration up to 24 Hours Post Dosing (AUC24h) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post-dose on Day 1
  The AUC24h is the area under the concentration versus time curve (AUC) from time of administration up to 24 hours post dosing.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post-dose on Day 1
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
AUC From Time 0 to Infinite Time (AUC[0-infinity]) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post-dose on Day 1
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Half-Life (t1/2) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post-dose on Day 1
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Clearance (CL/F) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post-dose on Day 1
  Total clearance of drug after extravascular administration, uncorrected for absolute bioavailability, calculated as: Dose (D)/AUC (0-infinity).
Apparent Volume of Distribution (Vd/F) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post-dose on Day 1
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Maximum Observed Concentration (Cmax) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 1
  Cmax is the maximum observed concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neuss, Germany